CLINICAL TRIAL: NCT00342017
Title: Immunological Consequences of Helminth and Mycobacterial Coinfection
Brief Title: The Effect of Parasitic Worm Infections on the Immune Response to Tuberculosis Bacteria
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901261; 01-I-N261
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-04

CONDITIONS: Intestinal Helminth Infection; Filarial Infection
Keywords: Filarial Infections; Helminths; Tuberculosis; Filarial Infection
MeSH Terms: conditions — Tuberculosis

SUMMARY:
This study, sponsored by the National Institutes of Health and the Tuberculosis Research Centre in Chennai, India, will examine how helminth and filarial infections affect the immune response to mycobacteria (the bacteria that causes tuberculosis). Helminths are parasitic worms that infect the gut, and filaria are worms that circulate in the blood and infect various tissues. The findings of this study may affect how tuberculosis is assessed in Chennai, where filarial and helminth infections are common in the population.

Patients between 6 and 65 years of age with helminth or filarial infections who do not have active tuberculosis, cancer, AIDS, or other immunosuppressive illness may be eligible for this study. Participants will be recruited from villages in the Chingleput District of Chennai, India.

Participants will complete a medical history and physical examination. They will have a blood test to determine red blood cell count and to detect filarial infection, a stool examination to detect helminth infection, and a tuberculin skin test for tuberculosis. Patients with a positive tuberculin test will be treated for tuberculosis and any filarial or helminth infections that may have been detected.

Patients whose tuberculin test is negative will be invited to participate in the second part of the study-to determine whether people with either filarial infections or helminth infections, or both, respond to tuberculosis bacteria in the same way as people who do not have these infections. Participants will undergo a review of their medical history, a physical examination, and a blood test to assess red blood cell levels and to look for evidence of filarial or helminth infection. They will then be randomly assigned to receive either albendazole and DEC (anti-helminth and anti-filarial drugs) or a placebo (look-alike tablets that do not contain an active ingredient). Two months later, patients will receive a second dose of the same tablets (placebo or active drug) they took previously, and after another 4 weeks they will be re-tested for tuberculosis. After 6 months (at the end of the study) all participants will receive anti-helminth and anti-filarial drugs and will have a repeat tuberculin skin test. Blood and stool samples will be collected twice in the 6-month period after the initial treatment to determine the levels of antibody against the parasites, to measure the level of infection with filaria, and to measure the level of red blood cells.

DETAILED DESCRIPTION:
To determine if preexisting intestinal helminth infection or filarial infection alters the immune response to mycobacterial antigens or the clinical expression of tuberculosis, this study proposes to assess the skin test reactivity to tuberculin (PPD) in a community in which intestinal helminth infection, filarial infection and tuberculosis co-exist. Once baseline data are obtained, all those who are PPD negative (but who harbor helminth parasites) will be randomized to receive either anthelminthics or placebo twice over a six week period. One and 4 months following the last dose, change in PPD status will be assessed as will the intestinal and filarial parasite burden. By assessing these changes, the influence of intestinal helminth or filarial infection on the cellular immune response to Mycobacterium tuberculosis can be determined.

ELIGIBILITY:
* INCLUSION CRITERIA:

Ages 6-65

Able to give informed consent (greater than 18 years)/parent's consent (less than 18 years) in case of children/young adults

Both sexes providing women are neither pregnant nor breastfeeding

Willingness to provide stool and blood for examination two times over a 6 month period

No known active tuberculosis, cancer, AIDS or other immunosuppressive illness

EXCLUSION CRITERIA:

Less than 6 years old or greater than 65 years old

Pregnant or breastfeeding by history

Known active tuberculosis, cancer, AIDS, other immunosuppressive illness. Active tuberculosis is defined as culture proven M. tuberculosis.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5200
Dates: Start 2002-05-20; Primary Completion 2008-09-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Tuberculosis Research Centre, Chennai, India

REFERENCES:
- [Background] Actor JK, Shirai M, Kullberg MC, Buller RM, Sher A, Berzofsky JA. Helminth infection results in decreased virus-specific CD8+ cytotoxic T-cell and Th1 cytokine responses as well as delayed virus clearance. Proc Natl Acad Sci U S A. 1993 Feb 1;90(3):948-52. doi: 10.1073/pnas.90.3.948. PMID 8094248
- [Background] Baily GV. Tuberculosis prevention Trial, Madras. Indian J Med Res. 1980 Jul;72 Suppl:1-74. No abstract available. PMID 7005086
- [Background] Bentwich Z, Weisman Z, Moroz C, Bar-Yehuda S, Kalinkovich A. Immune dysregulation in Ethiopian immigrants in Israel: relevance to helminth infections? Clin Exp Immunol. 1996 Feb;103(2):239-43. doi: 10.1046/j.1365-2249.1996.d01-612.x. PMID 8565306